CLINICAL TRIAL: NCT00346541
Title: Investigating the Genetic Basis of Glaucoma: Role of Polymorphisms in the IL-1 Gene Cluster
Brief Title: Role of Polymorphisms in the IL-1 Gene Cluster
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Other Study IDs: R423/18/2005
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2006-06-30 (Estimated); Status verified 2006-06

CONDITIONS: Glaucoma
Keywords: glaucoma; polymorphism, genetic
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Glaucoma, an optic neuropathy characterized by progressive visual field loss, is the leading cause of irreversible blindness worldwide. The condition has a substantial heritable basis, as illustrated by the numerous loci and genes identified to date, and the large proportion of patients having a family history.

Interleukin-1 (Il-1) is an important mediator of inflammation. There are 2 pro-inflammatory cytokines, Il-1 alpha and Il-1 beta. The genes encoding Il-1 are located within a 430kb region on chromosome 2q14.2. The role of Il-1 in glaucoma is a subject of recent interest. It has been shown that Il-1, produced endogenously by glaucomatous cells, inhibits the apoptotic response to oxidative stress, and Il-1 has also been reported to increase outflow facility by stimulating the _expression of matrix metalloproteinase enzymes, which in turn reduces extra cellular resistance. Recently, polymorphisms in Il-1 (particularly +3953T of the Il-1 β) were found to reduce the risk of primary open angle glaucoma. In this pilot study, we aim to investigate the role of Il-1 polymorphisms in both normal tension and high pressure glaucoma in our glaucoma patients. Both open and closed angle glaucoma will be studied. This is a pilot study of the role of immune system related polymorphisms and depending on the results, we may embark on a larger investigation of other immune genes in glaucoma

DETAILED DESCRIPTION:
Aims:

Primary objective: To investigate if polymorphisms in the Il-1 gene cluster are protective for glaucoma in Asian populations.

Secondary objective: To determine if there are differences in single nucleotide polymorphisms of the Il-1 gene cluster in normotensive glaucoma patients versus high-pressure glaucoma patients.

Background

The glaucomas are a group of heterogeneous optic neuropathies characterized by progressive loss of axons in the optic nerve. Based on WHO Global Data Bank on Blindness, glaucoma accounts for 5.1 million of the estimated 38 million blind in the world.1Glaucoma affects approximately 70 million people worldwide and is the leading cause of irreversible blindness in the world2. As the number of elderly in the world rapidly increases, glaucoma morbidity will rise, causing increased health care costs and economic burden. This has important public health implications for a condition in which visual loss, once established, cannot be reversed. The major risk factor in glaucoma is elevated intraocular pressure due to reduction in aqueous outflow.

Previous studies have shown that glaucoma is a major cause of visual morbidity in Singapore3-5. In a population based survey conducted on Chinese Singaporeans in the Tanjong Pagar district, the age-standardized prevalence of glaucoma was found to be 3.2% (95% confidence interval, 2.3-4.1) in the population 40 years and older.3

Glaucoma has a major genetic basis, estimated to account for a third (range 20 - 60%) of all glaucoma cases, 6-8 although a recent report suggests that this is an underestimate.9 Genetic heterogeneity is illustrated by the more than 15 loci and 7 glaucoma-causing genes identified to date, 10 including 2 genes identified for POAG.11-12 A diverse variety of genetic mechanisms have been found to induce open angle and developmental glaucomas and these include coding mutations, particularly in transcription factors, 13 altered gene dosage14 and dominant negative effects.15

Interleukin-1 is an important mediator of inflammation. There are 2 pro-inflammatory cytokines, Il-1 alpha and Il-1 beta. Both are produced by monocytes, macrophages and epithelial cells as host responses to tissue injury. The genes encoding Il-1 are located within a 430kb region on chromosome 2q14.216. Polymorphisms of the Il-1 gene cluster have been shown to alter protein _expression. Single nucleotide polymorphisms have been linked to other diseases such as pre-eclampsia among other medical conditions17.

_Expression of the endothelial leukocyte adhesion molecule-1 (ELAM-1) in trabecular meshwork cells has been identified to be a diagnostic marker of glaucoma18. _Expression of ELAM-1 is controlled by activation of Il-1 autocrine feedback loop, which is controlled through transcription factor NF-Kappa -Beta. It has been shown that Il-1 produced endogenously by glaucomatous cells inhibits the apoptotic response to oxidative stress18. Il-1 has also been reported to increase outflow facility by stimulating the _expression of matrix metalloproteinase enzymes, which in turn reduces extra cellular resistance19-22. The effect of Il-1 on the synthesis of Nitric oxide causing a relaxation in ciliary muscle tone may also be contributory in increasing aqueous outflow23.

Recently, Wang et al has shown that Il-1 variants result in increased secretion of Il-1 and thus reduces the risk of primary open angle glaucoma (POAG) 24. This was presented at the recent ARVO meeting 2005 in Florida, USA, under " New ideas in glaucoma". The group led by Dr Elizabeth Fini from Bascom Palmer Eye Institute, Miami, identified genetic variants (+3953T) of the Il-1 β, which is a protective factor against POAG. They assessed genomic DNA from 100 POAG patients and 104 normal controls in the Caucasian population over 40 years. The allele frequency of Il-1 Beta (+3953T) was significantly higher in normal controls than in the POAG group (28% versus 17%, p=0.01). They also found that the allele frequency of Il-1 alpha (-889T) was higher in normal controls than in the POAG group at borderline significance (39% versus 29%, p=0.06). This may prove to be significant with a larger sample size.

In this project, we hope to determine if polymorphisms in the Il-1 gene cluster found in the Caucasians are also protective for glaucoma patients in Asian populations. We also aim to determine if there are differences in the distribution of polymorphisms of the Il-1 gene cluster in normotensive glaucoma patients versus high-pressure glaucoma patients. Both primary angle closure and primary open angle glaucoma patients will be studied. The study will be the first to investigate such changes in PACG, a major cause of blindness in Asia, and considered to be an IOP-dependent disease. The study findings may have implications on the genetic basis of glaucoma, placing the focus on the role of the immune system in IOP response and glaucoma pathogenesis. This is a pilot study of the role of immune system related polymorphisms and depending on the results, we may embark on a larger investigation of the role of other immune genes in glaucoma.

Methods

Patient Recruitment:

At least 300 patients with primary glaucoma will be recruited in the study from glaucoma clinics at Singapore National Eye Centre. This will consist of PACG, POAG and NTG patients. There will be another 100 control patients with no clinical evidence of glaucoma recruited from the general clinics. Individuals with secondary angle closure and other ocular diseases will be excluded.

Patient assessment and examination Examination, of both eyes, will include best-corrected Snellen visual acuity, goniscopy, intraocular pressure measurement by Goldmann applanation tonometer, slit-lamp examination of the anterior segment, lens, vitreous and retina. In addition, a scanning laser ophthalmoscope, the Heidelberg retina tomograph (HRT, Heidelberg Engineering, Heidelberg, Germany) will be used to image the optic disc in all subjects. Global and segmental disc and cup areas will be analysed directly by means of HRT software (version 2.01b) using the standard reference plane. Rim area will be calculated by subtracting the cup area from the disc area. Glaucoma severity will be classified by global indices in the visual fields as well as by HRT neuroretinal rim area. Axial length will also be measured with the IOL-Master (Carl Zeiss Jena GmbH, Jena, Germany). 10 mls of blood will be obtained from each patient by venepuncture.

Standardized inclusion criteria for glaucoma will be used, which is the presence of glaucomatous optic neuropathy (defined as loss of neuroretinal rim with a cup:disc ratio of 0.7 or greater) with compatible visual field loss. PACG will be defined as the presence of at least 180 degrees of angle in which the trabecular meshwork is not visible on gonioscopy with the presence of glaucomatous optic neuropathy. POAG patients will have open angles on gonioscopy; POAG patients with a mean IOP without treatment that is consistently less than 21 mm Hg on diurnal testing will be classified as NTG.

DNA Preparation and Genotyping

Genomic DNA will be extracted from leukocytes of the peripheral blood using Nucleon DNA Extraction kits. The Il-1alpha (-889), Il-beta (-511), and Il-1beta (+3953) variants will be detected by specific polymerase chain reaction (PCR) (using primers in Table 1), followed by digestion with restriction enzyme digests as described in Table 1. Confirmation of polymorphisms would be carried out by direct sequencing.

The methodology is fairly straightforward and the lab work can be performed by Dr Alicia How (Registrar, SNEC) during her research session each week. Dr How has undergone basic molecular genetics lab training and will be supervised by Dr Aung Tin.

Table 1. Primer sequence, PCR condition and enzyme for the IL-1α (-889), IL-1β (-511), and IL-1β( +3953)

Polymorphism Primer sequence Annealing Temp (oC) Enzyme Expected DNA products (bp) IL-1alpha (-889) Forward 5'-GCATGCCATCACACCTAGTT-3' 58 Nco1 C:194 Reverse 5'-TTACATATGAGCCTTCCATG-3' T:178,16 IL-1beta (-511) Forward 5'-TGGCATTGATCTGGTTCATC-3' 60 Bsu36I, C:304 Reverse 5'-GTTTAGGAATCTTCCCACTT-3' T:190,114 IL-1beta (+3953) Forward 5'-GTTGTCATCAGACTTTGACC-3' 60 TaqI, C:135,114 Reverse 5'-TTCAGTTCATATGGACCAGA-3' T:249

ELIGIBILITY:
Inclusion Criteria:

* Standardized inclusion criteria for glaucoma will be used, which is the presence of glaucomatous optic neuropathy (defined as loss of neuroretinal rim with a cup:disc ratio of 0.7 or greater) with compatible visual field loss. PACG will be defined as the presence of at least 180 degrees of angle in which the trabecular meshwork is not visible on gonioscopy with the presence of glaucomatous optic neuropathy. POAG patients will have open angles on gonioscopy; POAG patients with a mean IOP without treatment that is consistently less than 21 mm Hg on diurnal testing will be classified as NTG.

There will be another 100 control patients with no clinical evidence of glaucoma recruited from the general clinics.

Exclusion Criteria:

* Individuals with secondary angle closure and other ocular diseases will be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Tin Aung, PHD, FRCS, Study Director — Singapore Eye Research Institute
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore